CLINICAL TRIAL: NCT01351805
Title: Vitamin D and Fish Oil for Autoimmune Disease, Inflammation and Knee Pain
Acronym: VITAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Karen H. Costenbader, Associate Physician, Brigham and Women's Hospital
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: R01AR059086 (NIH); R01AR059086 (NIH)
Record Dates: First submitted 2011-05-04; First posted 2011-05-11 (Estimated); Results first posted 2021-01-08 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Autoimmune Diseases; Systemic Inflammatory Process; Knee Pain Chronic; Osteoarthritis; Rheumatoid Arthritis
Keywords: vitamin D; omega-3 fatty acid; fish oil; prevention; trial; autoimmune disease; rheumatoid arthritis; psoriasis; systemic inflammation; Interleukin-6; C-reactive peptide; tumor necrosis factor; osteoarthritis
MeSH Terms: conditions — Autoimmune Diseases; Osteoarthritis; Arthritis, Rheumatoid; Psoriasis | interventions — Fish Oils; Eicosapentaenoic Acid; Docosahexaenoic Acids; Fatty Acids, Omega-3; Vitamin D; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Fish Oil (Experimental): Subjects will receive marine omega-3 fatty acids (465 mg of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA]).
  Interventions: Drug: Fish Oil; Other: placebo pill
- Vitamin D (Experimental): Subjects will receive vitamin D3 (cholecalciferol) 2000 IU a day.
  Interventions: Dietary Supplement: Vitamin D; Other: placebo pill
- placebo (Placebo Comparator): Subjects will receive placebo pill.
  Interventions: Other: placebo pill
- Vitamin D and Fish Oil (Experimental): Subjects will receive marine omega-3 fatty acids (465 mg of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA]).
  Interventions: Drug: Fish Oil; Dietary Supplement: Vitamin D

INTERVENTIONS:
Drug: Fish Oil — Subjects will receive marine omega-3 fatty acids (465 mg of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA]).
  Other Names: eicosapentaenoic acid (EPA); docosahexaenoic acid (DHA); marine fatty acids; omega-3 fatty acids; fish oils
  Arms: Fish Oil; Vitamin D and Fish Oil
Dietary Supplement: Vitamin D — Subjects will receive vitamin D3 (cholecalciferol) 2000 IU a day.
  Other Names: cholecalciferol; vitamin D3
  Arms: Vitamin D; Vitamin D and Fish Oil
Other: placebo pill — placebo
  Arms: Fish Oil; Vitamin D; placebo

SUMMARY:
The VITamin D and OmegA-3 TriaL (VITAL; NCT 01169259) is a randomized clinical trial in 25,871 U.S. men and women investigating whether taking daily dietary supplements of vitamin D3 (2000 IU) or omega-3 fatty acids (Omacor® fish oil, 1 gram) reduces the risk of developing cancer, heart disease, and stroke in people who do not have a prior history of these illnesses. This ancillary study is being conducted among VITAL participants and will examine whether vitamin D or fish oil have effects upon A) autoimmune disease incidence, B) biomarkers of systemic inflammation, and C) chronic knee pain. Blood samples at baseline and in follow-up will be collected in a randomly selected subcohort of 1500 individuals and analyzed for changes in biomarkers of systemic inflammation: C-reactive protein, interleukin-6, and tumor necrosis factor-receptor 2. Approximately 1300 individuals with chronic, frequent knee pain will be followed with annual questionnaires to evaluate the effects of the supplements on chronic knee pain.

ELIGIBILITY:
As for the parent trial, VITamin D and OmegA-3 TriaL (VITAL; NCT 01169259). Individuals with chronic, frequent knee pain at study baseline will be followed as a subcohort. Trial enrollment complete.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25871 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2018-11-10 (Actual); Study Completion 2025-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen H Costenbader, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Oakes EG, Vlasakov I, Kotler G, Bubes V, Mora S, Tatituri R, Cook NR, Manson JE, Costenbader KH. Joint effects of one year of marine omega-3 fatty acid supplementation and participant dietary fish intake upon circulating lipid mediators of inflammation resolution in a randomized controlled trial. Nutrition. 2024 Jul;123:112413. doi: 10.1016/j.nut.2024.112413. Epub 2024 Feb 28. PMID 38518540
- [Result] Costenbader KH, Cook NR, Lee IM, Hahn J, Walter J, Bubes V, Kotler G, Yang N, Friedman S, Alexander EK, Manson JE. Vitamin D and Marine n-3 Fatty Acids for Autoimmune Disease Prevention: Outcomes Two Years After Completion of a Double-Blind, Placebo-Controlled Trial. Arthritis Rheumatol. 2024 Jun;76(6):973-983. doi: 10.1002/art.42811. Epub 2024 Feb 20. PMID 38272846
- [Result] Costenbader KH, MacFarlane LA, Lee IM, Buring JE, Mora S, Bubes V, Kotler G, Camargo CA Jr, Manson JE, Cook NR. Effects of One Year of Vitamin D and Marine Omega-3 Fatty Acid Supplementation on Biomarkers of Systemic Inflammation in Older US Adults. Clin Chem. 2019 Dec;65(12):1508-1521. doi: 10.1373/clinchem.2019.306902. Epub 2019 Nov 7. PMID 31699704
- [Result] MacFarlane LA, Cook NR, Kim E, Lee IM, Iversen MD, Gordon D, Buring JE, Katz JN, Manson JE, Costenbader KH. The Effects of Vitamin D and Marine Omega-3 Fatty Acid Supplementation on Chronic Knee Pain in Older US Adults: Results From a Randomized Trial. Arthritis Rheumatol. 2020 Nov;72(11):1836-1844. doi: 10.1002/art.41416. Epub 2020 Oct 3. PMID 32583982
- [Result] Hahn J, Cook NR, Alexander EK, Friedman S, Walter J, Bubes V, Kotler G, Lee IM, Manson JE, Costenbader KH. Vitamin D and marine omega 3 fatty acid supplementation and incident autoimmune disease: VITAL randomized controlled trial. BMJ. 2022 Jan 26;376:e066452. doi: 10.1136/bmj-2021-066452. PMID 35082139
- See also: Welcome to the VITAL Study Website — http://www.vitalstudy.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From the 25871 VITAL participants, we identified 2 main subcohorts: A "systemic inflammation" subcohort of 1561 participants with sufficient blood biomarker assays, balanced by sex, and matched on blood draw season, and a second "knee pain" subcohort including 1,398 participants who returned one knee pain questionnaire and qualified at baseline. Both subcohorts are described below in their respective aims.
Pre-assignment Details: At 1 year, 95% of participants returned follow-up questionnaires, and approximately 90% were taking more than two-thirds of study pills (definition of compliance).
  Participants willing to provide a blood sample were sent a kit with consent form, supplies, and instructions to have blood drawn.
Groups:
- ACTIVE Vitamin D + ACTIVE Omega-3 Fatty Acids: ACTIVE Vitamin D = Vitamin D3, one 2000 IU capsule/day; ACTIVE Omega-3 Fatty Acids = Omacor, one 1-gram capsule/day. Each capsule of Omacor contains 840 milligrams of marine omega-3 fatty acids (465 mg of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA]).
- ACTIVE Vitamin D + PLACEBO Omega-3 Fatty Acids: ACTIVE Vitamin D = Vitamin D3, one 2000 IU capsule/day; PLACEBO Omega-3 Fatty Acids, one capsule/day
- PLACEBO Vitamin D + ACTIVE Omega-3 Fatty Acids: PLACEBO Vitamin D, one capsule/day; ACTIVE Omega-3 Fatty Acids = Omacor, one 1-gram capsule/day. Each capsule of Omacor contains 840 milligrams of marine omega-3 fatty acids (465 mg of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA]).
- PLACEBO Vitamin D + PLACEBO Omega-3 Fatty Acids: PLACEBO Vitamin D, one capsule/day; PLACEBO Omega-3 Fatty Acids, one capsule/day
Period: Overall Study
Arm/Group | ACTIVE Vitamin D + ACTIVE Omega-3 Fatty Acids | ACTIVE Vitamin D + PLACEBO Omega-3 Fatty Acids | PLACEBO Vitamin D + ACTIVE Omega-3 Fatty Acids | PLACEBO Vitamin D + PLACEBO Omega-3 Fatty Acids
Started | 6463 | 6464 | 6470 | 6474
Completed | 6463 | 6464 | 6470 | 6474
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: In this 2x2 factorial design trial, the primary analyses were: all active vitamin D vs. all placebo vitamin D and all active omega-3 fatty acids vs. all placebo omega-3 fatty acids.
Groups:
- Total: Total of all reporting groups
Arm/Group | ACTIVE Vitamin D + ACTIVE Omega-3 Fatty Acids | ACTIVE Vitamin D + PLACEBO Omega-3 Fatty Acids | PLACEBO Vitamin D + ACTIVE Omega-3 Fatty Acids | PLACEBO Vitamin D + PLACEBO Omega-3 Fatty Acids | Total
Number analyzed (Participants) | 6463 | 6464 | 6470 | 6474 | 25871
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2458 | 2462 | 2461 | 2467 | 9848
  >=65 years | 4005 | 4002 | 4009 | 4007 | 16023
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.1 (7.1) | 67.1 (7.0) | 67.2 (7.1) | 67.1 (7.1) | 67.1 (7.1)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 3276 | 3271 | 3271 | 3267 | 13085
  Male | 3187 | 3193 | 3199 | 3207 | 12786
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Race/Ethnicity measured using different categories in systemic inflammation versus knee pain subcohorts.
  Participants
    Non-Hispanic white | 4515 | 4498 | 4529 | 4504 | 18046
    African American | 1278 | 1275 | 1271 | 1282 | 5106
    Hispanic (not African American) | 246 | 270 | 245 | 252 | 1013
    Asian/Pacific Islander | 102 | 86 | 98 | 102 | 388
    Native American/ Alaskan Native | 62 | 56 | 58 | 52 | 228
    Other/ unknown | 126 | 133 | 123 | 141 | 523
Region of Enrollment [Number; unit: participants]
  United States | 6463 | 6464 | 6470 | 6474 | 25871

OUTCOME MEASURES:

1. Primary Outcome: Serum Levels of Biomarkers of Systemic Inflammation: Interleukin-6 (IL-6)
Description: In a subsample of the randomized trial population across the four arms, blood samples at baseline and in follow-up were collected and analyzed for changes in biomarkers of systemic inflammation: C-reactive protein (CRP), interleukin-6 (IL-6), and tumor necrosis factor-receptor 2 (TNFR2). We tested whether either or both supplements were associated with a decrease in the biomarkers of systemic inflammation (blood biomarker levels among those receiving supplements vs. placebo). We also tested whether there were interactions between the two supplements in their effects on changes in the IL-6 serum biomarker of systemic inflammation.
Time Frame: Baseline and 1 year
Population: Subsample of the VITAL trial participants at baseline and one year.
Measure: Geometric Mean (95% Confidence Interval); unit: pg/ml
Groups:
- Active Vitamin D: Vitamin D3, one 2000 IU capsule/day
- Placebo Vitamin D: Vitamin D placebo, one capsule/day
- Active n-3 FA: Omacor, one 1-g capsule/day. Each capsule of Omacor contains 840 mg of marine omega-3 fatty acids (465 mg of EPA + 375 mg of DHA).
- Placebo n-3 FA: Omega-3 fatty acids placebo, one capsule/day
Arm/Group | Active Vitamin D | Placebo Vitamin D | Active n-3 FA | Placebo n-3 FA
Number analyzed (Participants) | 784 | 777 | 784 | 777
pg/ml
  Baseline ln (IL-6) pg/ml, geometric mean (95% Cl) | 1.71 [1.65 to 1.78] | 1.68 [1.61 to 1.74] | 1.69 [1.63 to 1.75] | 1.70 [1.63 to 1.77]
  Year 1 ln (IL-6) pg/mL, geometric mean (95% CI) | 1.80 [1.73 to 1.87] | 1.63 [1.57 to 1.69] | 1.70 [1.64 to 1.77] | 1.72 [1.66 to 1.79]
Statistical Analysis 1: Comparison: Active Vitamin D vs Placebo Vitamin D; Geometric means of biomarker concentrations with 95% CIs were calculated for baseline and 1 year biomarkers (IL-6, TNFR2 and CRP) by treatment group (active vs. placebo vitamin D). Linear repeated measures models calculated the % change in means for each biomarker from baseline to year one and the overall effects of randomized treatments with 95% CIs; Test type: Other — Test of change from baseline as above; p = 0.02, as above — IL-6 from baseline to one year: overall % change= 8.19% (95%CI 1.52-15.31); p above adjusted for age, sex, race and n-3 fatty acid randomized treatment group; Percent change in geometric means = 8.19, 95% CI 2-sided [1.52 to 15.31]
Statistical Analysis 2: Comparison: Active n-3 FA vs Placebo n-3 FA; [analysis description as in outcome 1, analysis 1]; Test type: Other — Test of change from baseline as above; p = 0.97, as above — 4. IL-6 from baseline to one year: overall % change= -0.73% (95%CI -6.87 to 5.81); p above adjusted for age, sex, race and vitamin D randomized treatment group; Percent change in geometric means = -0.73, 95% CI 2-sided [-6.87 to 5.81]
Statistical Analysis 3: Comparison: Active Vitamin D vs Placebo Vitamin D vs Active n-3 FA vs Placebo n-3 FA; Test for interaction between effect of vitamin D and effect of omega-3 fatty acids on IL-6 change from baseline to 1 year; Test type: Superiority — Multiplicative interaction between strata based on linear models of ln biomarker from baseline to year 1,p for interaction between strata; p = 0.12, p for interaction — Test of multiplicative interaction between the effects of the two supplements

2. Primary Outcome: Serum Levels of Biomarkers of Systemic Inflammation: C-reactive Protein (CRP)
Description: In a subsample of the randomized trial population across the four arms, blood samples at baseline and in follow-up were collected and analyzed for changes in biomarkers of systemic inflammation: C-reactive protein (CRP), interleukin-6 (IL-6), and tumor necrosis factor-receptor 2 (TNFR2). We tested whether either or both supplements were associated with a decrease in the biomarkers of systemic inflammation (blood biomarker levels among those receiving supplements vs. placebo). We also tested whether there were interactions between the two supplements in their effects on changes in the CRP serum biomarker of systemic inflammation.
Time Frame: Baseline and 1 year
Population: Subsample of the VITAL trial participants at baseline and one year.
Measure: Geometric Mean (95% Confidence Interval); unit: mg/L
Arm/Group | Active Vitamin D | Placebo Vitamin D | Active n-3 FA | Placebo n-3 FA
Number analyzed (Participants) | 784 | 777 | 784 | 777
mg/L
  Baseline ln (hsCRP) mg/L, geometric mean (95% Cl) | 1.48 [1.40 to 1.57] | 1.51 [1.43 to 1.60] | 1.57 [1.49 to 1.66] | 1.43 [1.35 to 1.51]
  Year 1 ln (hsCRP) mg/L, geometric mean (95% CI) | 1.62 [1.53 to 1.71] | 1.54 [1.46 to 1.63] | 1.63 [1.54 to 1.72] | 1.53 [1.45 to 1.62]
Statistical Analysis 1: Comparison: Active Vitamin D vs Placebo Vitamin D; [analysis description as in outcome 1, analysis 1]; Test type: Other — Test of change from baseline as above; p = 0.16, as above — 3. HsCRP from baseline to one year: overall % change= 7.12% (95%CI -1.81-16.78); p above adjusted for age, sex, race and n-3 fatty acid randomized treatment group; Percent change in geometric means = 7.12, 95% CI 2-sided [-1.81 to 16.87]
Statistical Analysis 2: Comparison: Active n-3 FA vs Placebo n-3 FA; [analysis description as in outcome 1, analysis 1]; Test type: Other — Test of change from baseline as above; p = 0.44, as above — 6. HsCRP from baseline to one year: overall % change= -3.89% (95%CI -11.92-4.86); p above adjusted for age, sex, race and vitamin D randomized treatment group; Percent change in geometric means = -3.89, 95% CI 2-sided [-11.92 to 4.86]
Statistical Analysis 3: Comparison: Active Vitamin D vs Placebo Vitamin D vs Active n-3 FA vs Placebo n-3 FA; Test for multiplicative interaction between effect of vitamin D and effect of omega-3. based on linear models of ln biomarker from baseline to year 1; Test type: Superiority; p = 0.38, P for interaction

3. Primary Outcome: Serum Levels of Biomarkers of Systemic Inflammation: Tumor Necrosis Factor-receptor 2 (TNFR2)
Description: In a subsample of the randomized trial population across the four arms, blood samples at baseline and in follow-up were collected and analyzed for changes in biomarkers of systemic inflammation: C-reactive protein (CRP), interleukin-6 (IL-6), and tumor necrosis factor-receptor 2 (TNFR2). We tested whether either or both supplements were associated with a decrease in the biomarkers of systemic inflammation (blood biomarker levels among those receiving supplements vs. placebo). We also tested whether there were interactions between the two supplements in their effects on changes in the TNFR2 serum biomarker of systemic inflammation.
Time Frame: Baseline and 1 year
Population: Subsample of the VITAL trial participants at baseline and one year.
Measure: Geometric Mean (95% Confidence Interval); unit: pg/ml
Arm/Group | Active Vitamin D | Placebo Vitamin D | Active n-3 FA | Placebo n-3 FA
Number analyzed (Participants) | 784 | 777 | 784 | 777
pg/ml
  Baseline ln (TNFR2) pg/ml, geometric mean (95% Cl) | 2546.5 [2508.6 to 2584.9] | 2525.4 [2482.7 to 2568.9] | 2571.3 [2528.1 to 2615.2] | 2500.9 [2463.6 to 2538.8]
  Year 1 ln (TNFR2) pg/mL, geometric mean (95% CI) | 2604.7 [2565.2 to 2644.7] | 2567.9 [2523.9 to 2612.7] | 2605.3 [2561.4 to 2649.9] | 2567.3 [2527.7 to 2607.6]
Statistical Analysis 1: Comparison: Active Vitamin D vs Placebo Vitamin D; [analysis description as in outcome 1, analysis 1]; Test type: Other — Test of change from baseline as above; p = 0.57, as above — 2. TNFR2 from baseline to one year: overall % change= 0.63% (95%CI -1.03 to 2.31); p above adjusted for age, sex, race and n-3 fatty acid randomized treatment group; Percent change in geometric means = 0.63, 95% CI 2-sided [-1.03 to 2.31]
Statistical Analysis 2: Comparison: Active n-3 FA vs Placebo n-3 FA; [analysis description as in outcome 1, analysis 1]; Test type: Other — Test of change from baseline as above; p = 0.13, as above — 5. TNFR2 from baseline to one year: overall % change= -1.27% (95%CI -2.89 to 0.39); p above adjusted for age, sex, race and vitamin D randomized treatment group; Percent change in geometric means = -1.27, 95% CI 2-sided [-2.89 to 0.39]
Statistical Analysis 3: Comparison: Active Vitamin D vs Placebo Vitamin D vs Active n-3 FA vs Placebo n-3 FA; [analysis description as in outcome 2, analysis 3]; Test type: Superiority — Multiplicative interaction between strata based on linear models of ln biomarker from baseline to year 1 with p for interaction between strata; p = 0.74, P for interaction

4. Primary Outcome: Incident Autoimmune Diseases
Description: All participants were followed for the development of new autoimmune diseases, including, but not limited to, rheumatoid arthritis, psoriasis, autoimmune thyroid disease, inflammatory bowel disease and polymyalgia rheumatica. The primary endpoint was all incident autoimmune disease confirmed by extensive medical record review. Participants self-reported all incident autoimmune diseases from baseline through follow-up. We used Cox proportional hazards models to test the effects of vitamin D and n-3 fatty acids upon autoimmune disease incidence.
  We compared the separate main effects of vitamin D or n-3 fatty acid supplement assignment on AD incidence using Cox regression models. To account for randomization stratification and study design, we additionally adjusted for age, sex, self-reported race, and randomization to the other supplement. Person-time was counted until diagnosis of a new confirmed AD, death, or the end of the trial. We also test interactions between the two supplements
Time Frame: 5 years
Population: All participants in VITAL followed for the development of new autoimmune diseases, including, but not limited to, rheumatoid arthritis, psoriasis, autoimmune thyroid disease, inflammatory bowel disease and polymyalgia rheumatica. Categorized by vitamin D (active/placebo) and n-3 (active/placebo)
Measure: Count of Participants; unit: Participants
Arm/Group | Active Vitamin D | Placebo Vitamin D | Active n-3 FA | Placebo n-3 FA
Number analyzed (Participants) | 12927 | 12944 | 12933 | 12938
Participants | 123 | 155 | 130 | 148
Statistical Analysis 1: Comparison: Active Vitamin D vs Placebo Vitamin D; Test type: Other; p = 0.05, Regression, Cox; Cox Proportional Hazard = 0.78, 95% CI 2-sided [0.61 to 0.99]
Statistical Analysis 2: Comparison: Active n-3 FA vs Placebo n-3 FA; Test type: Superiority; p = 0.19, Regression, Cox; Cox Proportional Hazard = 0.85, 95% CI 2-sided [0.67 to 1.08]
Statistical Analysis 3: Comparison: Active Vitamin D vs Placebo Vitamin D vs Active n-3 FA vs Placebo n-3 FA; Test for multiplicative interaction between the effects of randomized treatment groups, vitamin D and n-3 fa on incidence of autoimmune disease; Test type: Superiority; p = 0.20, P for interaction; p multiplicative interaction between effects of vitamin D and n-3 fa supplements

5. Primary Outcome: Severity of Knee Pain in Subsample With Chronic, Frequent Knee Pain at Baseline- With n-3 FA & Vitamin D
Description: Western Ontario and McMaster University Osteoarthritis Index (WOMAC) Pain was the primary outcome on a scale of 0-100 with 100= worst pain.
  Subsample of VITAL participants with chronic, frequent knee pain at trial baseline were followed with annual WOMAC questionnaires to test for change in severity of chronic knee pain in those taking Omega-3 fish oil (n-3 FA) supplements compared to those taking placebo and for those taking Vitamin D supplements compared to those taking placebo. We tested whether n-3 FA supplements and Vitamin D are associated with reduced levels of WOMAC knee pain at the end of the trial (comparing knee pain outcomes in those receiving supplements to placebo). We will also test whether there were multiplicative interactions between the two supplements for the outcome of knee pain severity by WOMAC-Pain index
Time Frame: Baseline and 5 years
Population: Subsample of the VITAL trial who reported chronic frequent knee pain prior to randomization.
Measure: Mean (Standard Deviation); unit: WOMAC units on a scale
Groups:
- Active n-3 FA: Omacor, one 1-g capsule/day. Each capsule of Omacor contains 840 mg of marine omega-3 fatty acids (465 mg of EPA + 375 mg of DHA) + Vitamin D3, one 2000 IU capsule/day or Vitamin D placebo, one capsule/day
- Placebo n-3 FA: Omega-3 fatty acids placebo, one capsule/day + Vitamin D3, one 2000 IU capsule/day or Vitamin D placebo, one capsule/day
- Active Vitamin D: Vitamin D3, one 2000 IU capsule/day + Omega 3 Omacor fatty acid, 1-g capsule/day or Omega-3 fatty acid placebo
- Placebo Vitamin D: Placebo vitamin D3, one 2000 IU capsule/day + Omega 3 Omacor fatty acid, 1-g capsule/day or Omega-3 fatty acid placebo
Arm/Group | Active n-3 FA | Placebo n-3 FA | Active Vitamin D | Placebo Vitamin D
Number analyzed (Participants) | 595 | 626 | 591 | 630
WOMAC units on a scale
  Baseline mean WOMAC Pain | 36.5 (0.7) | 35.4 (0.7) | 35.4 (0.7) | 36.5 (0.7)
  Follow Up mean WOMAC pain | 33.6 (0.9) | 33.7 (0.9) | 32.7 (0.9) | 34.6 (0.9)
Statistical Analysis 1: Comparison: Active n-3 FA vs Placebo n-3 FA; Intention to treat analysis using a repeated measures model with unstructured variance to assess the effect of treatment arm on WOMAC Pain adjusting for age, sex, and the other treatment arm. The linear time by treatment interaction term assessed change in WOMAC Pain over time between participants randomized to treatment versus placebo; Test type: Other — We assessed the main effects of the treatment arms comparing all those randomized to omega-3 fatty acids or omega-3 fatty acid placebo, regardless of vitamin D randomization status; p = 0.77, Mixed Models Analysis — Repeated measures model with unstructured variance to assess effect of treatment on WOMAC Pain adjusting for age, sex, and other treatment. Linear time by treatment interaction term assessed change in WOMAC Pain over time in treatment vs placebo; Repeated measures model with censoring for total knee replacement
Statistical Analysis 2: Comparison: Active Vitamin D vs Placebo Vitamin D; [analysis description as in outcome 5, analysis 1]; Test type: Other — We assessed the main effects of the treatment arms comparing all those randomized to vitamin D or vitamin D placebo, regardless of omega-3 fatty acid randomization status; p = 0.41, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]; Linear time by treatment interaction (comparing change in WOMAC pain over time in two randomized groups); We assessed for effect modification between vitamin D and N-3 FA and tested for other pre-specified interactions. We again used a repeated measures model with censoring for TKR. We adjusted for age, sex and N-3 FA treatment arm (in analyses in which N-3 FA treatment arm was not investigated as a potential modifier)
Statistical Analysis 3: Comparison: Active n-3 FA vs Placebo n-3 FA vs Placebo Vitamin D; Active n3fa vs placebo n3fa among those on placebo vitamin D; Test type: Other — Linear regression - WOMAC pain over time mean (Standard error - SE). Differences in WOMAC pain scores in stratified groups; p = 0.42, Regression, Linear; Mean Difference (Net) = -1.5, Standard Error of Mean 1.9
Statistical Analysis 4: Comparison: Placebo n-3 FA vs Active Vitamin D vs Placebo Vitamin D; Vitamin D vs. vitamin D placebo among those on placebo omega-3 fatty acids- stratified analyses; Test type: Other — [test comment as in outcome 5, analysis 3]; p = 0.18, Regression, Linear; Mean Difference (Net) = -2.5, Standard Error of Mean 1.8
Statistical Analysis 5: Comparison: Active n-3 FA vs Placebo n-3 FA vs Active Vitamin D; Omega-3 fatty acids vs. omega-3 fatty acids placebo among those on active vitamin D; Test type: Other — Linear regression - WOMAC pain over time mean (Standard error - SE). Report only in final year. Differences in WOMAC pain scores in cross-classified groups; p = 0.84, Regression, Linear; Mean Difference (Net) = 0.39, Standard Error of Mean 1.89
Statistical Analysis 6: Comparison: Active n-3 FA vs Placebo n-3 FA vs Placebo Vitamin D; Omega-3 fatty acids vs. omega-3 fatty acids placebo among those on placebo vitamin D; Test type: Other — [test comment as in outcome 5, analysis 5]; p = 0.76, Regression, Linear; Mean Difference (Net) = -0.55, Standard Error of Mean 1.80

6. Secondary Outcome: Incident Autoimmune Disease
Description: Development of new autoimmune disease through observational follow-up after trial termination.
Time Frame: extension of follow-up through 2 years post trial closure, up to 7 years
Population: Baseline enrolled populations
Measure: Count of Participants; unit: Participants
Groups:
- Active Vitamin D: 2000IU vitamin D3 orally per day
- Placebo Vitamin D; Placebo n-3 FA: placebo pill: placebo
- Active n-3 FA: marine omega-3 fatty acids (465 mg of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA]) orally per day
Arm/Group | Active Vitamin D | Placebo Vitamin D | Active n-3 FA | Placebo n-3 FA
Number analyzed (Participants) | 12927 | 12944 | 12933 | 12938
Participants | 255 | 259 | 234 | 280
Statistical Analysis 1: Comparison: Active Vitamin D vs Placebo Vitamin D vs Active n-3 FA vs Placebo n-3 FA; HR for incident autoimmune disease in intervention groups vs. placebo (ref=1.0) using Cox models with 95% confidence intervals; Test type: Superiority; p < 0.05, Regression, Cox — HR with 95%CI; Hazard Ratio (HR) = 1.0

ADVERSE EVENTS:
Time Frame: 5 years
Description: Vit D Monitored safety cond'ns: hypercalcemia, kidney stones, parathyroid disease, kidney failure or dialysis; Other symptoms, side effects: GI bleeding, easy bruising; stomach upset or pain; nausea; constipation, diarrhea, skin rash
  Omega-3 FA Monitored safety cond'ns: GI bleeding; blood in urine; easy bruising; freq nosebleeds; kidney failure or dialysis; Other symptoms, side effects: stomach upset or pain; nausea; constipation; diarrhea; skin rash; bad taste in mouth; increased burping
Groups:
- Active Vitamin D/ Active Omega-3 Fatty Acids: Vitamin D3, one 2000 IU capsule/day
  Omacor, one 1-g capsule/day. Each capsule of Omacor contains 840 mg of marine omega-3 fatty acids (465 mg of EPA + 375 mg of DHA).
- Active Vitamin D/ Active Omega-3 Placebo: Vitamin D3, one 2000 IU capsule/day
  Omega-3 fatty acids placebo, one capsule/day
- Active Omega-3 Fatty Acids, Placebo Vitamin D: Omacor, one 1-g capsule/day. Each capsule of Omacor contains 840 mg of marine omega-3 fatty acids (465 mg of EPA + 375 mg of DHA).
  Vitamin D placebo, one capsule/day
- Omega-3 Fatty Acids Placebo/ Placebo Vitamin D: Omega-3 fatty acids placebo, one capsule/day
  Vitamin D placebo, one capsule/day
Arm/Group | Active Vitamin D/ Active Omega-3 Fatty Acids | Active Vitamin D/ Active Omega-3 Placebo | Active Omega-3 Fatty Acids, Placebo Vitamin D | Omega-3 Fatty Acids Placebo/ Placebo Vitamin D
All-Cause Mortality (participants affected / at risk) | 241/6463 | 244/6464 | 252/6470 | 241/6474
Serious Adverse Events (participants affected / at risk) | 791/6463 | 782/6464 | 822/6470 | 837/6474
Other Adverse Events (participants affected / at risk) | 5101/6463 | 5027/6464 | 5037/6470 | 5101/6474
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Vitamin D/ Active Omega-3 Fatty Acids (N=6463) | Active Vitamin D/ Active Omega-3 Placebo (N=6464) | Active Omega-3 Fatty Acids, Placebo Vitamin D (N=6470) | Omega-3 Fatty Acids Placebo/ Placebo Vitamin D (N=6474)
Gastrointestinal bleeding (Blood and lymphatic system disorders) | 170 | 171 | 200 | 203
Hypercalcemia (Endocrine disorders) | 77 | 70 | 74 | 69
Invasive cancer of any type (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 408 | 385 | 412 | 412 — Total cancer = invasive cancer of any type
Death from cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 75 | 79 | 93 | 94
Breast cancer (in women) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 60 | 64 | 57 | 65
Prostate cancer (in men) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 109 | 83 | 110 | 109
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 28 | 23 | 26 | 21
Major cardiovascular event (Vascular disorders) | 186 | 210 | 200 | 209 — Major cardiovascular event = a composite endpoint of myocardial infarction, stroke, and death from cardiovascular causes
Myocardial infarction (Vascular disorders) | 72 | 97 | 73 | 103
Stroke (Vascular disorders) | 66 | 75 | 82 | 67
Death from cardiovascular causes (Vascular disorders) | 74 | 78 | 68 | 70
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Vitamin D/ Active Omega-3 Fatty Acids (N=6463) | Active Vitamin D/ Active Omega-3 Placebo (N=6464) | Active Omega-3 Fatty Acids, Placebo Vitamin D (N=6470) | Omega-3 Fatty Acids Placebo/ Placebo Vitamin D (N=6474)
Easy bruising (Blood and lymphatic system disorders) | 1737 | 1697 | 1706 | 1702
Frequent nosebleeds (Blood and lymphatic system disorders) | 224 | 242 | 241 | 249
Blood in urine (Blood and lymphatic system disorders) | 469 | 442 | 450 | 432
Parathyroid condition (Endocrine disorders) | 24 | 26 | 28 | 34 — Parathyroid condition = hyperparathyroidism or hypoparathyroidism
Stomach upset or pain (Gastrointestinal disorders) | 2439 | 2421 | 2448 | 2422
Nausea (Gastrointestinal disorders) | 1748 | 1771 | 1810 | 1779
Constipation (Gastrointestinal disorders) | 2567 | 2566 | 2617 | 2545
Diarrhea (Gastrointestinal disorders) | 2781 | 2730 | 2818 | 2850
Increased burping (Gastrointestinal disorders) | 1107 | 1061 | 1110 | 1097
Bad taste in mouth (General disorders) | 1109 | 1086 | 1131 | 1159
Kidney stones (Renal and urinary disorders) | 233 | 244 | 197 | 229
Kidney failure or dialysis (Renal and urinary disorders) | 42 | 43 | 43 | 45
Skin rash (Skin and subcutaneous tissue disorders) | 1629 | 1639 | 1702 | 1728

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2009-11-09): https://cdn.clinicaltrials.gov/large-docs/05/NCT01351805/Prot_SAP_000.pdf